CLINICAL TRIAL: NCT01445691
Title: A Multicenter Phase II Study of 5-Aminolevulinic Acid (ALA) to Enhance Visualization and Resection of Newly Diagnosed or Recurrent Malignant Gliomas
Brief Title: More Complete Removal of Malignant Brain Tumors by Fluorescence-Guided Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Constantinos Hadjipanayis (Other)
Collaborators: NX PharmaGen (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Constantinos Hadjipanayis, Professor and Chair, Neurosurgery, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 15-2034; WCI1999-11 (Other: Other); R01CA176659 (NIH); R21CA186169 (NIH); IRB00051663 (Other: Emory University)
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Benign Neoplasms, Brain; Brain Cancer; Brain Neoplasms, Benign; Brain Neoplasms, Malignant; Brain Tumor, Primary; Brain Tumor, Recurrent; Brain Tumors; Intracranial Neoplasms; Neoplasms, Brain; Neoplasms, Intracranial; Primary Brain Neoplasms; Primary Malignant Brain Neoplasms; Primary Malignant Brain Tumors; Gliomas; Glioblastoma
Keywords: Benign Neoplasms, Brain; Brain Cancer; Brain Neoplasms, Benign; Brain Neoplasms, Malignant; Brain Tumor, Primary; Brain Tumor, Recurrent; Brain Tumors; Intracranial Neoplasms; Neoplasms, Brain; Neoplasms, Intracranial; Primary Brain Neoplasms; Primary Malignant Brain Neoplasms; Primary Malignant Brain Tumors; Gliomas; Glioblastoma; Surgery; 5-ALA; Aminolevulinic acid; Fluorescence
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5-ALA (Gliolan) (Experimental): Fluorescent substance to help visualize and remove as much tumor as possible without harming healthy tissue.
  Interventions: Drug: 5-ALA (Gliolan)

INTERVENTIONS:
Drug: 5-ALA (Gliolan) — 20 mg/kg administered once 3-5 hours prior to surgery
  Other Names: 5-ALA; Aminolevulinic acid; Gliolan

SUMMARY:
The purpose of this study is to determine the safety and utility of 5-aminolevulinic acid (ALA) for identifying your tumor during surgery. 5-ALA is not FDA approved at this time. When the investigators remove the tumor from your brain, it is important that they remove all of the tumor and not remove parts of normal brain. Sometimes this can be difficult because the tumor can look like normal brain. In some brain tumors, 5-ALA can make the tumors glow red under blue light. This may make it easier for your doctor to take out all of the tumor from your brain. The purpose of this study is to:

* Make sure that 5-ALA helps the doctor remove more of the tumor.
* Make sure 5-ALA does not cause any side effects.

If you do not want to participate in this study, your doctor(s) will still do their best to remove all of the tumor in your brain. Whether or not you join this study will not change your treatment for your brain tumor.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinically documented primary brain tumor for which resection is clinically indicated. Individuals with suspected newly diagnosed or recurrent malignant gliomas will be considered eligible for the study. The anticipated histology at resection should include: Anaplastic astrocytoma (10002224), Anaplastic ependymoma, Anaplastic oligodendroglioma, Astrocytoma malignant NOS (10003572), Glioblastoma (10018336), Glioblastoma multiforme (10018337), or Gliosarcoma (10018340).
* Prior therapy is not a consideration in protocol entry.
* Age 18-80.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%).
* Life expectancy is not a consideration for protocol entry.
* Subjects must have normal organ and marrow function as defined below:

  * Leukocytes ≥ 3,000/mL
  * Platelets ≥ 100,000/mL
  * Total bilirubin below upper limit of normal
  * Aspartate aminotransferase (AST) (SGOT)/alanine aminotransferase (ALT) (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Creatinine below upper limit of normal OR
  * Creatinine clearance ≥ 60 mL/min/1.73 m² for patients with creatinine levels above institutional normal
* The effects of aminolevulinic acid (ALA) on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A pregnancy test will be performed for all women of childbearing ability prior to surgery. Women who are pregnant will be excluded from the trial.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Tumors of or involving the midline, basal ganglia, or brain stem as assessed by MRI.
* Subjects may not be receiving any experimental therapies.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to aminolevulinic acid (ALA). Patients should refrain from use of other potential phototoxic substances (e.g. tetracyclines, sulfonamides,fluoroquinolones, hypericin extracts) for 72 hours.
* Personal or family history of porphyrias.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Pregnant women are excluded from this study because aminolevulinic acid (ALA) is of unknown teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with aminolevulinic acid (ALA), breastfeeding should be discontinued if the mother is treated with aminolevulinic acid (ALA).
* Women who are pregnant will be excluded from the trial.
* Prior history of GI perforation, diverticulitis, and/or peptic ulcer disease.
* Inclusion of women and minorities: both men and women and members of all ethnic groups are eligible for this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Radicality of Brain Tumor Resection | Within the first 48 hours after surgery

SECONDARY OUTCOMES:
Progression-free survival every 3 months after surgery | Every 3 months until tumor progression on MRI

CONTACTS AND LOCATIONS:
Overall Officials: Costas Hadjipanayis, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (6):
- United States (6):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri